CLINICAL TRIAL: NCT03902990
Title: Effects of Dual Task Training And Treadmill Training on Physical and Cognitive Functions in Patients With Parkinson Disease
Brief Title: The Effect of Dual Tasking on Physical and Cognitive Functions in Patients With Parkinson Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Tugce Kocamal, Assistant Doctor, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20181443
Record Dates: First submitted 2019-04-03; First posted 2019-04-04 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Parkinson Disease
Keywords: dual task, treadmill, cognitive rehabilitation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: In this prospective, randomized, controlled, double-blinded study the patients were randomized to three groups as; dual-task group, single-task group and control group. All of the patients were scheduled on standard exercise programme. The patients in dual-task group received treadmill training with cognitive tasks and the patients in single-task group received treadmill training alone in addition to standard exercise programme. The training was scheduled as 30 minute sessions under supervision of a specialist, three times in a week for four weeks.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dual task (Experimental): Treadmill training + cognitive tasks + standard exercise programme
  Interventions: Other: Dual task; Other: Treadmill Training; Other: Standard exercise programme
- Single task (Active Comparator): Treadmill training + standard exercise programme
  Interventions: Other: Treadmill Training; Other: Standard exercise programme
- Control (Active Comparator): Standard exercise programme
  Interventions: Other: Standard exercise programme

INTERVENTIONS:
Other: Dual task — The patients in the dual task group received cognitive tasks during treadmill training sessions.
  Arms: Dual task
Other: Treadmill Training — Standard treadmill training
  Arms: Dual task; Single task
Other: Standard exercise programme — Standard exercise programme for Parkinson Disease

SUMMARY:
The ability of performing multi-tasking procedures is impaired in patients with Parkinson's disease. In this study, our goal was to detect the effects of dual-task training with treadmill training on walking and balance and to compare its effects on quality of life, cognitive functions and risk of fall, to treadmill training alone.

ELIGIBILITY:
Inclusion Criteria:

The patients with Idiopathic Parkinson Disease on medication who has

* Hoehn-Yahr 1-3
* Mini Mental Test score 20 and above
* Functional Ambulation Category 2 and above
* No changes in medication in last 3 months
* No rehabilitation programme in last 3 months

Exclusion Criteria:

* Diagnosis of Parkinsonism other than Idiopathic Parkinson Disease
* Global aphasia
* Severe cognitive dysfunction
* Other neurologic/orthopedic diseases
* Limiting cardiovascular or pulmonary disease
* Visual impairment
* Hearing loss

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
10MWT | 12 weeks
  10 Meter Walk Test on comfortable speed
10MWT with cognitive tasks | 12 weeks
  10 Meter Walk Test with cognitive tasks
MoCA | 12 weeks
  Montreal Cognitive Assessment
TUG | 12 weeks
  Timed Up and Go Test

SECONDARY OUTCOMES:
PDQ-39 | 12 weeks
  Parkinson Disease Questionnaire 39
FES-I | 12 weeks
  To evaluate fear of falling, all patients filled the Falls Efficacy Scale-International (FES-I). A series of 16 questions assesses the respondent's fear of falling for a range of ADLs. Each question was rated on a four-point scale.
Stroop Test | 12 weeks
  Cognitive assessment for executive functions
FOGQ | 12 weeks
  Freezing of Gait Questionnaire
Falls Diary | 4 weeks
  Falls account

CONTACTS AND LOCATIONS:
Overall Officials: Ayse Yaliman, Prof, Study Director — Istanbul University Istanbul Faculty of Medicine Physical Medicine and Rehabilitation; Ekin Ilke Sen, MD, Study Director — Istanbul University Istanbul Faculty of Medicine Physical Medicine and Rehabilitation
Locations (1):
- Istanbul University Istanbul Faculty of Medicine Department of Physical Medicine and Rehabilitation, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No